CLINICAL TRIAL: NCT06854757
Title: Families Left Behind: Addressing Prolonged Grief and Substance Use Disorders Among People Bereaved by Drug Overdose Deaths
Brief Title: Families Left Behind
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Stanford University (Other); Peer Support Community Partners (Unknown)
Responsible Party: Principal Investigator, Alison Athey, Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-N0522
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Grief; Grief Disorder, Prolonged; Overdose Accidental; Substance Use Disorders
Keywords: overdose; grief; bereavement; prolonged grief disorder
MeSH Terms: conditions — Prolonged Grief Disorder; Substance-Related Disorders; Drug Overdose | interventions — Rivers

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized controlled trial (RCT) of peer grief support plus enhanced care as usual vs. enhanced care as usual only (i.e., parallel interventional study model).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer grief support + enhanced care as usual (Experimental): Participants in this arm will be matched with a peer grief support specialist who will provide support that aligns with the RIVER process model developed by Peer Community Support Partners. They will also receive a psychoeducational booklet and a list of local grief support resources (i.e., the enhanced care as usual condition).
  Interventions: Behavioral: RIVER; Behavioral: Enhanced care as usual
- Enhanced care as usual (Active Comparator): Participants will receive a psychoeducational booklet and a list of local grief support resources.
  Interventions: Behavioral: Enhanced care as usual

INTERVENTIONS:
Behavioral: RIVER — RIVER is a peer grief support process intervention developed by Peer Support Community Partners.
  Arms: Peer grief support + enhanced care as usual
Behavioral: Enhanced care as usual — The enhanced care as usual condition involves a psychoeducational booklet developed by What's Your Grief, as well as a list of local grief resources.

SUMMARY:
The United States is facing unprecedented rates of drug overdose deaths, profoundly impacting millions of families who are left to navigate their grief. Those bereaved by overdose experience a unique form of grief characterized by feelings of guilt, shame, and blame, which can worsen their suffering and deter them from seeking help. Individuals coping with overdose loss often endure more severe health consequences compared to those grieving non-drug related deaths, including prolonged grief disorder, substance use disorders, PTSD, depression, and suicidal thoughts. Moreover, bereaved individuals, particularly those with a history of substance use, may engage in risky behaviors as a means of coping, further exacerbating the risk of overdose and mortality within this vulnerable population. Peer grief support interventions have emerged as a promising approach to assist those experiencing such losses. To combat these outcomes, we are collaborating with Peer Community Support Partners (PSCP) in a novel practice-research partnership to implement the RIVER peer grief support model. Though RIVER has shown success in community settings, it has yet to be rigorously evaluated. In a three-aim approach, this study aims to assess the effectiveness of the RIVER model while also enhancing and engaging grievers with support resources via medical examiner offices (MEOs), which routinely contact families during death investigations. This research represents a pivotal advancement in addressing the needs of the overlooked bereaved community, aligning with the NIH's Helping to End Addiction Long-term (HEAL) initiative to develop effective strategies against the opioid crisis. Together, community engagement and rigorous research efforts aim to enhance support for those affected by the tragedy of drug overdose.

ELIGIBILITY:
Inclusion Criteria:

* people who lost a loved one to an unintentional drug overdose death within the past year
* age 18 and older
* fluently understand English or Spanish
* have the capacity to give consent (e.g., excluding those with severe cognitive impairment, those in active psychosis, and those with developmental disabilities).

Exclusion Criteria:

* people who need hospitalization for psychiatric symptoms or substance use disorders. (Note, people who use drugs but who do not require hospitalization will be included.)
* people have active suicidal ideation
* people who lost someone to a drug overdose death more than one year ago
* people who lost someone to a drug overdose death that was suicidal in nature or of undetermined intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Participant Grief Symptoms | Baseline, 3-month follow up, 6-month follow up, and 12-month follow up
  Brief Grief Questionnaire; evaluates the presence of prolonged grief
Participant Avoidance of Grief Reminders | Baseline, 3-month follow up, 6-month follow up, and 12-month follow up
  Grief-Related Avoidance Questionnaire (GRAQ); evaluating the presence and extent of avoidance behaviors due to feelings of grief
Participant Bereavement Coping Strategies | Baseline, 3-month follow up, 6-month follow up, and 12-month follow up
  Coping Assessment for Bereavement (CABLE); evaluating what coping strategies are being utilized and at what frequency
Participant Acceptance of the Loss | Baseline, 3-month follow up, 6-month follow up, and 12-month follow up
  Typical Beliefs Questionnaire (TBQ); evaluating the presence of maladaptive cognitions related to complicated grief
Participant Perceived Connectedness | Baseline, 3-month follow up, 6-month follow up, and 12-month follow up
  Continuing Bonds Scale; assessing the extent to which the participant feels bonded to the descendent

SECONDARY OUTCOMES:
Participant Substance Use | Baseline, 3-month follow up, 6-month follow up, and 12-month follow up
  Tobacco, Alcohol, Prescription Medications, and Other Substances Tool (TAPS); assessing the presence and frequency of past 30-day substance use
Participant Depression Severity | Baseline, 3-month follow up, 6-month follow up, and 12-month follow up
  Beck Depression Inventory (BDI); evaluating the presence and severity of depressive symptoms
Participant Posttraumatic Stress Symptoms | Baseline, 3-month follow up, 6-month follow up, and 12-month follow up
  Posttraumatic Stress Disorder Checklist (PCL-5); evaluating the severity of symptoms associated with posttraumatic stress disorder
Participant Physical Pain Severity | Baseline, 3-month follow up, 6-month follow up, and 12-month follow up
  PEG; evaluating the intensity and interference of physical pain on daily life and well-being

CONTACTS AND LOCATIONS:
Overall Officials: Alison Athey, PhD, Principal Investigator — RAND; Karen Osilla, PhD, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - Jefferson County Coroner/Medical Examiner's Office, Birmingham, Alabama
  - San Diego County Medical Examiner Office, San Diego, California
  - Connecticut Office of the Chief Medical Examiner, Farmington, Connecticut
  - Peer Support Community Partners, Watertown, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared by following NIH HEAL Data Sharing Policies.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Osilla KC, Watkins KE, Lord T, Lord G, Cook F, Nameth K, Kim JP, Hawkins W, Athey A. Study protocol for a randomized trial examining a peer grief support approach for people grieving drug overdose deaths. Res Sq [Preprint]. 2025 Aug 21:rs.3.rs-6959900. doi: 10.21203/rs.3.rs-6959900/v1. PMID 40894007